CLINICAL TRIAL: NCT02961686
Title: Quality of Life and Sexuality in Patients Treated With Radical Radiotherapy for Prostate Cancer
Brief Title: Quality of Life and Sexuality in Patients With Prostate Cancer
Status: Withdrawn | Type: Observational
Why Stopped: None patient was enrolled
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Medical Doctor, Istituto Clinico Humanitas
Other Study IDs: 1635
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with prostate cancer: Patients affected by prostate cancer and treated with a multidisciplinary approach that comprise exclusive radiotherapy, psychological and andrologic evaluation.
  Interventions: Radiation: Patients affected by prostate cancer

INTERVENTIONS:
Radiation: Patients affected by prostate cancer — Patients affected by prostate cancer and treated with a multidisciplinary approach: it includes exclusive radiotherapy, psychological and andrologic evaluation.

SUMMARY:
The trial is to describe quality of life in patients affected by prostate cancer treated with exclusive radiotherapy and submitted to psychological and andrologic evaluation.

DETAILED DESCRIPTION:
This trial is to describe quality of life and sexuality in patients with prostate cancer treated with exclusive radiotherapy. Descriptive analysis of baseline characteristics will be performed by using appropriate summary measures for continous and categorical data. Analysis of variation over time of FACT scores will be conducted by means of ANOVA analysis for repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years.
* Histologically-proven of prostate cancer
* Indication to radical radiotherapy on prostate/ prostate + seminal vesicles / prostate + seminal vesicles + pelvic lymph nodes
* Informed consent

Exclusion Criteria:

* Other coexisting malignancies, uncontrolled intercurrent illness, active infectious processes, and exudative, bloody, or cytologically malignant effusions excluded patients from the trial.
* Previous surgery for prostate cancer, severe cardiac or vascular pathology
* Other major surgery in the preceding year or currently undergoing psychiatric care or psychological counseling.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Quality of life measurement | 2.5 years
  Evaluation of the quality of life with FACT-P test in patient affected by prostate cancer treated with exclusive radiotherapy and submitted to psychological and andrologic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Franzese, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No